CLINICAL TRIAL: NCT03373435
Title: A Phase 2, Multicenter, Randomized, Single-Blind, Placebo-Controlled Cross-over Study to Assess the Efficacy and Safety of Exendin 9-39 in Patients With Postbariatric Hypoglycemia
Brief Title: Safety and Efficacy of Exendin 9-39 in Patients With Postbariatric Hypoglycemia
Acronym: PREVENT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eiger BioPharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: EIG-EXD-001
Record Dates: First submitted 2017-11-27; First posted 2017-12-14 (Actual); Results first posted 2022-06-28 (Actual); Last update posted 2022-07-18 (Actual); Status verified 2022-06

CONDITIONS: Postbariatric Hypoglycemia
MeSH Terms: interventions — exendin (9-39)

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment Group 1 (Experimental): patients will receive two dose regimens of exendin 9-39 and one placebo
  Interventions: Drug: exendin 9-39; Other: Placebo
- Treatment Group 2 (Experimental): patients will receive two dose regimens of exendin 9-39 and one placebo (in a different sequence than Treatment Group 1)
  Interventions: Drug: exendin 9-39; Other: Placebo

INTERVENTIONS:
Drug: exendin 9-39 — Exendin 9-39 is a competitive antagonist of GLP-1 at its receptor.
  Other Names: Avexitide
Other: Placebo — Placebo solution is identical to the active drug product except for the absence of the active ingredient, Exendin 9-39.

SUMMARY:
This clinical study will evaluate whether taking an investigational drug called exendin 9-39 is safe, well-tolerated, and helps to prevent low blood sugar in people who have had bariatric surgery and later develop a rare condition called postbariatric hypoglycemia (PBH).

DETAILED DESCRIPTION:
This is a Phase 2, multicenter, randomized, single-blind, placebo-controlled cross-over study in patients with refractory PBH.

Participants will be randomized and assigned in a 1:1 ratio to one of two treatment arms. All participants will receive 2 dosing regimens of exendin 9-39 and matching placebo self-administered via subcutaneous (SC) injection.

Participants will undergo in-clinic mixed meal tolerance test (MMTT) provocation with concomitant blood draws and symptom assessments.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) of up to 40 kg/m2
* Roux-en-Y gastric bypass (RYGB) surgery performed ≥12 months prior
* Diagnosis of PBH
* At least 2 episodes during screening 2-week run-in phase of severe hypoglycemia

Exclusion Criteria:

* Other cause of endogenous hyperinsulinism other than PBH
* Metabolic or bariatric surgical procedure other than RYGB
* History of non-RYGB upper GI surgery
* Use of agents that may interfere with glucose metabolism

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-03-19 (Actual); Primary Completion 2019-01-30 (Actual); Study Completion 2019-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Colleen Craig, MD, Study Director — Eiger BioPharmaceuticals, Inc
Locations (5):
- United States (5):
  - Stanford University, Palo Alto, California
  - University of Colorado, Denver, Aurora, Colorado
  - Johns Hopkins University, Baltimore, Maryland
  - Duke Early Phase Clinical Research, Durham, North Carolina
  - University of Wisconsin, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Craig CM, Lawler HM, Lee CJE, Tan M, Davis DB, Tong J, Glodowski M, Rogowitz E, Karaman R, McLaughlin TL, Porter L. PREVENT: A Randomized, Placebo-controlled Crossover Trial of Avexitide for Treatment of Postbariatric Hypoglycemia. J Clin Endocrinol Metab. 2021 Jul 13;106(8):e3235-e3248. doi: 10.1210/clinem/dgab103. PMID 33616643

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Group 1: Placebo first, then exendin 9-39 30 mg BID, then exendin 9-39 60 mg QD
  exendin 9-39: Exendin 9-39 is a competitive antagonist of glucagon-like peptide-1 (GLP-1) at its receptor.
  Placebo: Placebo solution is identical to the active drug product except for the absence of the active ingredient, Exendin 9-39.
- Treatment Group 2: Placebo first, then exendin 9-39 60 mg QD, then exendin 9-39 30 mg BID
  exendin 9-39: Exendin 9-39 is a competitive antagonist of GLP-1 at its receptor.
  Placebo: Placebo solution is identical to the active drug product except for the absence of the active ingredient, Exendin 9-39.
Period: Treatment Period 1 (14 Days)
Arm/Group | Treatment Group 1 | Treatment Group 2
Started | 8 | 10
Completed | 8 | 10
Not Completed | 0 | 0
Period: Treatment Period 2 (14 Days)
Arm/Group | Treatment Group 1 | Treatment Group 2
Started | 8 | 10
Completed | 8 | 10
Not Completed | 0 | 0
Period: Treatment Period 3 (14 Days)
Arm/Group | Treatment Group 1 | Treatment Group 2
Started | 8 | 10
Completed | 8 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Treatment Group 1 (Placebo, Exendin 9-39 30 mg BID, Exendin 9-39 60 mg QD): Placebo, exendin 9-39 30 mg BID, exendin 9-39 60 mg QD
  exendin 9-39: Exendin 9-39 is a competitive antagonist of GLP-1 at its receptor.
  Placebo: Placebo solution is identical to the active drug product except for the absence of the active ingredient, Exendin 9-39.
- Treatment Group 2 (Placebo, Exendin 9-39 60 mg QD, Exendin 9-39 30 mg BID): Placebo, exendin 9-39 60 mg QD, exendin 9-39 30 mg BID
  exendin 9-39: Exendin 9-39 is a competitive antagonist of GLP-1 at its receptor.
  Placebo: Placebo solution is identical to the active drug product except for the absence of the active ingredient, Exendin 9-39.
- Total: Total of all reporting groups
Arm/Group | Treatment Group 1 (Placebo, Exendin 9-39 30 mg BID, Exendin 9-39 60 mg QD) | Treatment Group 2 (Placebo, Exendin 9-39 60 mg QD, Exendin 9-39 30 mg BID) | Total
Number analyzed (Participants) | 8 | 10 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 10 | 18
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 10 | 18
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 7 | 10 | 17
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Weight [Mean (Standard Deviation); unit: kilograms] | 81.6 (7.3) | 81.0 (16.1) | 81.23 (12.6)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 30.0 (3.1) | 29.3 (4.9) | 29.6 (4.1)

OUTCOME MEASURES:

1. Primary Outcome: Postprandial Glucose Nadir
Description: Plasma glucose nadir occurring within 3 hours of mixed-meal tolerance testing (MMTT)
Time Frame: 3 hours following a liquid meal
Population: Analysis population are both treatment group 1 and treatment group 2. One participant was excluded from the efficacy analysis due to major protocol deviation.
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- Avexitide 30 mg BID: patients (treatment group 1 + treatment 2) received 30 mg twice a day
- Avexitide 60 mg QD: patients (treatment group 1 + treatment group 2)) receive 60 mg once a day.
- Placebo: Patients received placebo in treatment period 1 (initial 14 days) in the study.
Arm/Group | Avexitide 30 mg BID | Avexitide 60 mg QD | Placebo
Number analyzed (Participants) | 17 | 17 | 17
mg/dL | 57.1 (16.5) | 59.2 (16.1) | 47.1 (12.7)

ADVERSE EVENTS:
Time Frame: 3 Months
Description: Patients were evaluated and questioned to identify adverse events during the course of the study by the Investigator.
Groups:
- Avexitide 60 mg QD: patients (treatment group 1 + treatment group 2)) received 60 mg once a day.
Arm/Group | Avexitide 30 mg BID | Avexitide 60 mg QD | Placebo
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18 | 1/18 | 0/18
Other Adverse Events (participants affected / at risk) | 3/18 | 9/18 | 14/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Avexitide 30 mg BID (N=18) | Avexitide 60 mg QD (N=18) | Placebo (N=18)
presyncope (Nervous system disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Avexitide 30 mg BID (N=18) | Avexitide 60 mg QD (N=18) | Placebo (N=18)
Injection site bruising (General disorders) | 0 | 1 | 7
Headache (Nervous system disorders) | 1 | 1 | 4
Nausea (Gastrointestinal disorders) | 2 | 3 | 4
Dizziness (Nervous system disorders) | 0 | 1 | 1
Injection site pain (General disorders) | 0 | 1 | 1
Migraine (Nervous system disorders) | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-31): https://cdn.clinicaltrials.gov/large-docs/35/NCT03373435/Prot_SAP_000.pdf